CLINICAL TRIAL: NCT00615368
Title: The Effect of Intravenous Erythropoietin Treatment on Cognition During Hypoglycemia in Patients With Type 1 Diabetes.
Brief Title: Treatment With Erythropoietin and Cognition During Hypoglycaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: Maastricht University Medical Center (Other); Rigshospitalet, Denmark (Other); Steno Diabetes Center Copenhagen (Other); Erasmus Medical Center (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Peter Lommer Kristensen, MD, Hillerod Hospital, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-185; 2007-005651-41 (EudraCT Number); H-A-2007-0116 (Other: The Regional Committee on Biomedical Research Ethics)
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Type 1 diabetes; Hypoglycaemia; Cognitive function; Erythropoietin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Isotonic NaCl, intravenously injection
  Interventions: Drug: Isotonic NaCl (Placebo)
- Active (Experimental): Epoetin alfa, injected
  Interventions: Drug: Epoetin alfa

INTERVENTIONS:
Drug: Epoetin alfa — 1 (one) intravenously injection of 40.000 IU epoetin alfa 6 days before induction of experimental hypoglycemia.
  Other Names: Eprex
  Arms: Active
Drug: Isotonic NaCl (Placebo) — 1 ml. of isotonic NaCl is intravenously injected 6 days before induction of experimental hypoglycaemia
  Arms: Placebo

SUMMARY:
The purpose of the trial is to determine if erythropoietin (EPO) can enhance cognitive function during hypoglycaemia in patients with type 1 diabetes.

Patients with type 1 diabetes will receive one injection of EPO. Hypoglycaemia will be induced 6 days after. Before (1 hour), during and after (1 hour) hypoglycaemia, the cognitive function will be measured.

DETAILED DESCRIPTION:
Experimental protocol 6 days before hypoglycemic clamp subjects attended the clinic, and information about demography, lifestyle and clinical characteristics was collected. A physical examination with focus on possible thromboembolic disease was performed. Blood pressure was measured twice after 10 min rest in a sitting position. Measures of peripheral and autonomic neuropathy were assessed and a 12-lead electrocardiogram (ECG) was visually assessed. State of hypoglycemia awareness was classified according to Pedersen-Bjergaard et al [22]. The frequencies of episodes of mild and severe hypoglycemia in the preceding week were recorded in a questionnaire. A sensor for continuous glucose monitoring (CGM) was mounted (Guardian® REAL-time, Medtronic Minimed, Northridge, USA). Hereafter, the subject was re-introduced to the experimental protocol and cognitive tests were trained twice to avoid a learning effect during the experiments. Finally, study medication was injected intravenously over four minutes. Subjects were instructed to live and eat as they used to do, to avoid any rigorous exercise, use of alcohol and psychoactive drugs, for the next week. Calibration of the CGM was done by the patient with the blood glucose meter CONTOUR® LINK (Bayer Health Care, Leverkusen, Germany).

3 days before experiment A new CGM sensor was inserted and a hypoglycemia alarm was activated. Because the CGM glucose value is delayed approximately 10 min compared to plasma glucose the alarm-point was set to 4.5 mmol/l. CGM glucose profiles for the last three days were downloaded to check if any insulin dosage changes should be done to decrease the risk of hypoglycemia until the experiment 3 days later. Finally, the subjects trained the cognitive function tests again.

Day of experiment Subjects arrived at 8.00 a.m. in the laboratory after an overnight fast. Data from the CGM were downloaded. If hypoglycemia, defined by at least two consecutive CGM values below 3.5 mmol/l or one self-monitored blood glucose value below 3.5 mmol/l, had occurred during the preceding night, the experiment was postponed for at least 14 days. This was the case at one occasion. CGM warned the participants about decreasing blood glucose during the night before the experiment at three occasions before it actually occurred. In these cases the participants were instructed to eat a standardized meal of 10 grams of glucose and 35 g of dark bread. No participants had a CGM glucose > 20 mmol/l during the night before the experiments.

The subject was introduced to the experimental setting and was equipped as follows: 1) One antecubital intravenous line for infusion of insulin and glucose and one line as distally as possible for blood sampling. Thereafter, the hand and arm were placed on and under heated pads to arterialize venous blood; 2) EEG (electroencephalography) cap, two ear lobe references and two precordial ECG leads connected to a digital EEG recorder (Cadwell, Kennewick, Washington, USA); 3) an automatic blood pressure unit (UA787, A&D Medical, Abingdon, UK). Subsequently, subjects trained the cognitive tests.

The experiment was carried out in a cyclic manner with a total of three identical cycles: A baseline cycle (euglycemia), a hypoglycemic cycle and a recovery cycle (euglycemia). In the start of each cycle arterialized venous blood was drawn. Subsequently, hypoglycemic symptoms were assessed followed by measurement of blood pressure and pulse rate. Hereafter, evaluation of cognitive function was done with the California Cognitive Assessment Package (CALCAP), a trail making test and the Stroop test. All cognitive testing was conducted in the same sequence by the same person (PLK). At the end of each cycle, 5 min of EEG recording was done with eyes closed. Finally, arterialized venous blood was drawn again.

Hypoglycemic clamp procedure Short-acting human insulin (Actrapid®, Novo Nordisk, Bagsværd, Denmark) mixed with heparinized plasma from the patient and isotonic saline was infused at a rate of 1.0 mU x kg body weight-1 x min-1. Capillary blood glucose was measured bedside every 5 min and adjusted with a variable infusion of 20% glucose. The hypoglycemic target was 2.0 - 2.2 mmol/l. During the euglycemic cycles the target was 5.0 mmol/l.

Hypoglycemia symptom scoring Hypoglycemic symptoms were assessed by the The Edinburgh Hypoglycemia Scale, which is a questionnaire developed for experimentally induced hypoglycemia in which subjects must indicate the severity of 13 pre-defined hypoglycemic symptoms on a scale from one to seven [23].

Cognitive function tests California Cognitive Assessment Package (CALCAP) The Danish version of the Mini CALCAP test (E.N Miller, California Cognitive Assessment Package, Norland Software, Los Angeles, 1990) runs on a computer screen and consists of two different reaction time tasks with different complexity: 1) a choice reaction task (RT1) with reaction to a specific number (seven) and 2) a choice reaction task (RT2) with reaction to two identical numbers in a sequence (shifting numbers). The latter test is a 1-back task and includes the use of sustained attention/working memory.

Trail making test The trail making test is a test attention and executive function [24]. We used trail 5 of the Comprehensive Trail-Making Test (Pro-ed, Austin, Texas, USA), which is organized like the original trail making test, part B, developed in 1949, and added distracter circles [24]. In this test the subject must connect circled numbers and letters in alternating sequence (e.g. 1-A-2-B-3-C…). The time to finish the test was measured in seconds.

Stroop Color and Word Test This test measures selective attention and cognitive flexibility [25]. A Danish version of the standardized version by Golden [26] was used according to the test-manual. The test consists of three pages, each having 100 items presented in 5 columns. On the first page the words "red", "green" and "blue" are printed in black and arranged randomly. On the second page "XXXX" is printed in red, green or blue and arranged randomly. On the last page words from the word page are printed in non-matching colors from the color page. On the first and the second page the subject is supposed to read loud the color of the items. On the word-color-page the subject must read the color of the ink for each item. Number of items during a 45 second period is recorded. Raw scores are presented.

Neurophysiological tests Electroencephalography (EEG) A neurophysiologist specialized in clinical EEG reading (TWK) analyzed the EEG data. Continuous 20-channel EEG was recorded. Data were filtered by a first order 0.53 Hz low cut filter and a first order 70 Hz high cut filter. All data were visually inspected in a linked earlobe reference montage. For each subject the electrode giving the best representation of the dominant activity was chosen for power spectral analysis, which was performed using fast fourier transformation (FFT) on 2.5 sec epochs (giving 0.4 Hz resolution in the FFT power spectrum). If a peak in the power spectrum could be identified in the range 4-13 Hz, it was extracted as representative for the dominant frequency.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Hypoglycaemia unawareness
* 2 or more episodes of hypoglycaemia in the last 12 months
* Age >18 år
* Duration of diabetes > 5 år
* Weight > 50 kg
* No pregnancy
* Informed consent

Exclusion Criteria:

* Pregnancy
* Heart failure (NYHA 2-4)
* Ischaemic heart disease
* Epilepsy
* Venous thromboembolic disease
* Thrombocytosis
* Beta receptor antagonists
* Disturbance of vision
* History of stroke
* History of erythropoietin treatment
* Plasma-creatinin > 100 umol/l (male)or 88 umol/l (female)
* Plasma-haemoglobin < 7,0 or > 11 mmol/l at time of inclusion
* Operation with blood loss within the last 6 weeks
* Cancer
* Treated with ciclosporin
* Suspicion of non-compliance with protocol
* Conditions incompatible with participation - e.g. safety considerations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cognitive function | At baseline, during hypoglycemia and after hypoglycemia

SECONDARY OUTCOMES:
Hypoglycaemic counter regulatory symptoms | At baseline, during hypoglycemia and after hypoglycemia
Hypoglycemic hormonal response | At baseline, during hypoglycemia and after hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Kristensen, MD, Principal Investigator — Hillerod Hospital, Denmark
Locations (1):
- Hillerød Hospital, Hillerød, Hillerød, Denmark

REFERENCES:
- [Derived] Kristensen PL, Pedersen-Bjergaard U, Kjaer TW, Olsen NV, Dela F, Holst JJ, Faber J, Tarnow L, Thorsteinsson B. Influence of erythropoietin on cognitive performance during experimental hypoglycemia in patients with type 1 diabetes mellitus: a randomized cross-over trial. PLoS One. 2013;8(4):e59672. doi: 10.1371/journal.pone.0059672. Epub 2013 Apr 5. PMID 23577069